CLINICAL TRIAL: NCT00102310
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel Group, Dose Ranging Study of YM443 in Subjects With Functional Dyspepsia
Brief Title: YM443 in Subjects With Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 443-CL-008
Record Dates: First submitted 2005-01-26; First posted 2005-01-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Indigestion; Nausea
Keywords: Nausea; Indigestion; Bloating; Functional Dyspepsia; Fullness after Meals
MeSH Terms: conditions — Dyspepsia; Nausea

INTERVENTIONS:
Drug: YM443

SUMMARY:
The primary objective of this study will be to characterize the dose response profile of YM443 in subjects with functional dyspepsia (FD) to enable the selection of doses for the Phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in English.
* Written informed consent has been obtained.
* 18-75 years of age on the day the Informed Consent Form is signed.
* Men or women.
* Females, not pregnant, lactating or likely to become pregnant.
* Abdominal ultrasound and/or upper endoscopy findings that are judged as not clinically significant by the Investigator during Screening or within 4 weeks prior to Screening.
* Symptoms of FD at Visits 1 and 4 as defined by Rome II criteria.
* Subjects with a positive H. pylori breath test at Screening may be included in the study.
* Subjects with pH-metry results at Screening indicative of reflux may be included in the study.
* ECG, vital signs, and laboratory results that are judged as not clinically significant by the Investigator during Screening.

Exclusion Criteria:

* Significant renal, hepatic, bilirubin, cardiovascular, pulmonary, endocrine, metabolic, hematological, neurologic, or gastrointestinal (other than the one being studied) condition.
* Subjects with diabetes mellitus are to be excluded.
* Congenital or acquired long QT syndrome, or uncontrolled arrhythmias.
* Prior surgery on the luminal GI tract.
* History of any major psychiatric disorder, current depression or anxiety, alcohol abuse, or substance abuse in the last 2 years.
* Any evidence or treatment for malignancy (with the exception of basal cell carcinoma) within the last 5 years.
* Confirmed structural gastrointestinal disease.
* Predominant symptoms of irritable bowel syndrome (IBS) (Rome II criteria) or gastroesophageal reflux disease (GERD) assessed at Visit 1 or 4.
* Female subjects who are pregnant, lactating, or are likely to become pregnant during the study.
* Males and females of child-bearing potential must be abstinent or agree to use contraceptive regimens throughout the study.
* Any history or condition which, in the opinion of the Investigator, makes the subject unsuitable for any of the procedures used during this study or would not allow for safe completion of the study.
* Known hypersensitivity to gastroprokinetics or proton pump inhibitors.
* Use of anti-ulcer medications, antacid/acid suppression medications, gastroprokinetics, aspirin (>325 mg daily), other NSAIDs, antibiotics, and other medications that effect the GI system within 2 weeks prior to Screening. Must be able to stay off these medications during the study, except for proton pump inhibitors (PPIs) administered during the PPI Run-in Period.
* Required use of concomitant medications known to adversely interact with other gastroprokinetic agents or proton pump inhibitors.
* H. pylori eradication therapy (PPIs, antibiotics, bismuth preparations) in the 2 weeks prior to the upper endoscopy.
* Treatment for H. pylori required during the study.
* Subject has received an investigational drug within 30 days or 10 half-lives, which ever is longer, or participated in more than 3 clinical studies within 12 months, prior to Visit 1.
* Previous treatment with YM443.
* Employees of the Yamanouchi Group or CROs involved in the study.
* More than one subject per household to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2004-03-10 (Actual); Primary Completion 2006-03-11 (Actual); Study Completion 2006-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — APUS
Locations (59):
- United States (59):
  - Dr. Suresh Karne, Huntsville, Alabama
  - James Thrasher, MD, Little Rock, Arkansas
  - Dr. Dennis Riff, Anaheim, California
  - Dr. Peter Winkle, Cypress, California
  - Dr. Ramin Farsad, Encinitas, California
  - Dr. Prahalad Jajodia, Fresno, California
  - Dr. Gurmej Dhillon, Fresno, California
  - Dr. Steven Duckor, Orange, California
  - Dr. Theodor Feinstat, Roseville, California
  - Scott Levenson, MD, San Carlos, California
  - Dr. Michael Bennett, San Diego, California
  - Dr. William Snape, San Francisco, California
  - Dr. Abbass Shafii, Colorado Springs, Colorado
  - Dr. Julio Salcedo, Washington D.C., District of Columbia
  - Dr. Daniel Maico, Gainesville, Florida
  - Dr. Simon Behar, Hialeah, Florida
  - Wayne Schonfeld, MD, Hollywood, Florida
  - Dr. Stephen Palte, Atlanta, Georgia
  - Dr. Nathan Segall, Atlanta, Georgia
  - Azazuddin Ahmed, MD, Oak Brook, Illinois
  - Brian Covey, MD, Dubuque, Iowa
  - Dr. Richard McCallum, Kansas City, Kansas
  - Robert Braun, MD, Topeka, Kansas
  - Carroll Steinfeld, MD, Madisonville, Kentucky
  - David Dulitz, MD, Metairie, Louisiana
  - Dr. Bal Raj Bhandari, Monroe, Louisiana
  - Dr. Robert Hardi, Chevy Chase, Maryland
  - Dr. Braden Kuo, Boston, Massachusetts
  - Dr. Robert Lustig, Bridgewater, New Jersey
  - Dr. Rejendra Prasad Gupta, Trenton, New Jersey
  - Dr. Vitaly Fishbein, West Orange, New Jersey
  - Dr. Wieslaw Ignatowicz, Brooklyn, New York
  - Dr. Eugene Bonapace, Great Neck, New York
  - Dr. James Grendell, Mineola, New York
  - Dr. William Harlan, Asheville, North Carolina
  - Dr. John Poulos, Fayetteville, North Carolina
  - Dr. Peter Eweje, Jacksonville, North Carolina
  - Dr. Charles Barish, Raleigh, North Carolina
  - Dr. William Gramley, Wilmington, North Carolina
  - Dr. Robert Kindel, Cincinnati, Ohio
  - Dr. Gregory Cooper, Cleveland, Ohio
  - Dr. Gary Falk, Cleveland, Ohio
  - Dr. Michael Grossman, Oklahoma City, Oklahoma
  - Michael Mirhej, MD, Eugene, Oregon
  - Dr. Nayan Shah, Eynon, Pennsylvania
  - Dr. Robert Fisher, Philadelphia, Pennsylvania
  - Dr. Cynthia Strout, Mt. Pleasant, South Carolina
  - Robert Smith, MD, Saluda, South Carolina
  - Dr. Richard Krause, Chattanooga, Tennessee
  - Dr. Mark Swaim, Jackson, Tennessee
  - George James, MD, Nashville, Tennessee
  - Dr. Ronald Pruitt, Nashville, Tennessee
  - Dr. James Race, Dallas, Texas
  - Sardar Khan, MD, Houston, Texas
  - Ralph Alhalel, MD, McAllen, Texas
  - Dr. Daniel Pambianco, Charlottesville, Virginia
  - Dr. Mark Ringold, Christiansburg, Virginia
  - Vinod Rustgi, MD, Fairfax, Virginia
  - Dr. Michael Schmalz, Milwaukee, Wisconsin

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=65